CLINICAL TRIAL: NCT00606320
Title: A Multicenter, Investigative Study of the Safety and Efficacy of Extended Administration of Aripiprazole in Combination With Mood Stabilizer for the Treatment of Patients With Bipolar Disorder Experiencing a Manic or Mixed Episode
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-06-005
Record Dates: First submitted 2008-01-19; First posted 2008-02-01 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — oral, 24mg(4 tablets)/day
  Other Names: OPC-14597

SUMMARY:
To assess the safety and efficacy of long-term administration of aripiprazole by performing extended administration of aripiprazole in combination with mood stabilizer (lithium or valproate) in an unblinded manner to those patients who completed the preceding multicenter, double-blind, placebo-controlled, parallel group-comparison trial of aripiprazole in patients with bipolar disorder experiencing a manic or mixed episode (Study 031-06-003, hereafter "Study 003") but whose condition worsened or remained unchanged or who discontinued Study 003 between Day 14 and Day 21 due to lack of drug efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Trial subjects will be men and women of age 18 or above and below the age of 65 who will not be turning 65 during the trial.
* Subjects have the ability to understand and to provide informed consent to the examination, observation, and evaluation processes specified in this protocol, and have signed the informed consent form based on a full understanding of the trial.
* Subjects who meet DSM-IV-TR criteria for manic or mixed episodes and have been diagnosed as having "296.4x Bipolar I Disorder in which the most recent episode was manic" or "296.6x Bipolar I Disorder in which the most recent episode was mixed"
* Subjects who were enrolled in and have completed or withdrawn from Study 003 and who meet the following criteria

  * Subjects who show exacerbation of condition or no change in condition: Those subjects who completed Study 003, and whose score for CGI-BP Change from preceding phase (mania) on Day 21 (completion of Study 003) was between 5 (Minimally worse) and 7 (Very much worse) (subjects showing exacerbation of condition), or whose score was 4 (No change) (subjects showing no change in condition)
  * Subjects who discontinued due to lack of drug efficacy: Those subjects who discontinued Study 003 between Day 14 and Day 21, for whom the reason of withdrawal was lack of drug efficacy, and whose score for CGI-BP Change from preceding phase (mania) was between 5 (Minimally worse) and 7 (Very much worse)

Exclusion Criteria:

* Subjects presenting with a clinical picture and/or history that is consistent with a DSM-IV-TR diagnosis of:

  * Delirium, dementia, amnestic disorder, or other cognitive disorders
  * Schizophrenia or other psychotic disorder
  * Personality disorder
* Subjects with psychotic symptoms that are clearly due to another general medical condition or direct physiological effects of a substance
* Subjects who represent a significant risk of committing suicide
* Subjects known to have a complication of allergy to aripiprazole, other quinolinone-skeleton compounds, lithium, or valproate
* Subjects with a complication of neuroleptic malignant syndrome
* Subjects in a state of physical exhaustion accompanied by such conditions as dehydration or malnutrition
* Subjects with a complication of paralytic ileus
* Subjects with a complication of organic brain disorder or convulsive disorder, such as epilepsy
* Subjects with a complication of diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Department of Clinical Research and Development, Division of New Product Evaluation and Development
Locations (12):
- Hong Kong, China
- Japan (9):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Hokuriku Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region
- Seoul, South Korea
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazple: Patients who had completed the preceding study but whose condition worsened or remained unchanged or who discontinued the preceding study on Day 14 to Day 21 due to lack of drug efficacy were the target.
  Subjects were administered 24, 12, or 30mg/day of aripiprazole once daily for 154 days in an unblinded manner. Subjects were also administered mood stabilizer concomitantly for 154 days.
Period: Overall Study
Arm/Group | Aripiprazple
Started | 59
Completed | 22
Not Completed | 37
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 7
Not completed — Protocol Violation | 8
Not completed — Withdrawal by Subject | 10
Not completed — Progression to depressive phase | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Population(FAS)：Excluding the following subjects from the randomized subjects:
  * 3 subjects with GCP violation
  * 1 subject whose post dose efficacy were not available
Groups:
- Arupiprazole: Patients who had completed the preceding study but whose condition worsened or remained unchanged or who discontinued the preceding study on Day 14 to Day 21 due to lack of drug efficacy were the target.
  Subjects were administered 24, 12, or 30mg/day of aripiprazole once daily for 154 days in an unblinded manner. Subjects were also administered mood stabilizer concomitantly for 154 days.
Arm/Group | Arupiprazole
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (12.45)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 52
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 27
Region of Enrollment [Number; unit: participants]
  Taiwan | 5
  China | 17
  Japan | 11
  Malaysia | 6
  Indonesia | 4
  Philippines | 12

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: YMRS is composed of 11 evaluation items with 5 rating levels each. Items rated on a scale of 0 to 4 (comprising 5 rating levels of one point each) are 1) levated mood, 2) increased motor activity/energy, 3) sexual interest, 4) sleep, 7) language-thought disorder, 10) appearance, and 11) insight. Items rated on a scale of 0 to 8 (comprising 5 rating levels of two points each) are 5) irritability, 6) speech (rate and amount), 8) content, and 9) disruptive-aggressive behavior. YMRS ranges from 0 (best possible outcome) to 60 (worst possible outcome). Using LOCF datasets, descriptive statistics of actual values for changes of YMRS total scores from baseline (Day 1 of preceding study) to endpoint (Day 154) was calculated.
Time Frame: baseline (Day 1 of preceding study), Day 154 or at discontinuation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Aripiprazple
Number analyzed (Participants) | 55
scores on a scale | -18.3 (12.71)

2. Secondary Outcome: Clinical Global Impression - Bipolar Version (CGI-BP) Severity of Illness (Mania)
Description: CGI-BP severity of illness is a scale for overall evaluation of the severity of bipolar disorder; it comprises 3 components-mania, depression, and overall bipolar illness. CGI-BP severity of illness score (mania) ranges form 1 (normal, not ill) to 7 (very severely ill).
  Using LOCF datasets, descriptive statistics of actual values for change of CGI-BP severity of illness score (mania) from baseline (Day 1 of preceding study) to endpoint (Day 154) was calculated for each treatment group.
Time Frame: Baseline (Day 1 of preceding study) , Day 154 or at discontinuation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Aripiprazple
Number analyzed (Participants) | 55
scores on a scale | -2.4 (1.76)

ADVERSE EVENTS:
Time Frame: 22 weeks
Groups:
- Aripiprazole: Patients who had completed the preceding study but whose condition worsened or remained unchanged or who discontinued the preceding study on Day 14 to Day 21 due to lack of drug efficacy were the target.
Arm/Group | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 2/56
Other Adverse Events (participants affected / at risk) | 37/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=56)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=56)
Constipation (Gastrointestinal disorders) | 4 (8)
Salivary Hypersecretion (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 3 (3)
Nasopharyngitis (Infections and infestations) | 5 (5)
Weight Increased (Investigations) | 16 (16)
Alanine Aminotransferase Increased (Investigations) | 4 (4)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (3)
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 4 (4)
Akathisia (Nervous system disorders) | 12 (13)
Tremor (Nervous system disorders) | 10 (14)
Somnolence (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 5 (6)
Dystonia (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No